CLINICAL TRIAL: NCT05853757
Title: A Proof of Science/Concept Clinical Study With a Single-arm, Single-Blind to Evaluate Safety, Efficacy, and In-use Tolerability of Herbal Supplement in Healthy Adult Human Subjects Having Difficulty to Fall Asleep.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Herbal Supplement in Adult Human Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Vedistry Private Limited (Unknown)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator-Medical Director, NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NB230006-VPL
Record Dates: First submitted 2023-04-05; First posted 2023-05-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Difficulty in Sleep Initiation
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Proof of science/concept, Single-arm, Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zzowin Nutra Tablet (Experimental): Zzowin Nutra Tablet contains Melatonin, Tagar, L-theanine, L-Tryptophan, vitamin B6, Iron, Zinc, and Magnesium. which is helpful to provide deep, calm, and restful sleep.
  Interventions: Drug: Zzowin Nutra Tablet

INTERVENTIONS:
Drug: Zzowin Nutra Tablet — 1 Tablet daily half an hour before going to bed
  Other Names: Herbal Supplement

SUMMARY:
A proof of science/concept clinical study with single-arm, single-blind, to evaluate safety, efficacy and in-use tolerability study of Herbal Supplement in adult human subjects having difficulty in falling asleep.

A total of up to 32 subject will be enrolled to get 30 completed subject in the study.

DETAILED DESCRIPTION:
A sufficient number of adult subjects with an age group of 18 - 65 years old will be recruited/enrolled.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day -07): Screening within 7 days from Day 01
* Visit 02 (Day 01): Enrolment Day
* Visit 03 (Day 15): End of treatment
* Visit 04 (Day 30): Telephonic follow-up Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be telephonically contacted by recruiting department prior to the enrolment visit. Subjects will be instructed during screening (prior to enrolment) have to fill up the sleep diary before enrolment.

Assessment of safety and efficacy parameters will be done before test treatment usage on Day 1, and will be compared with after test treatment usage on Day 15 (+2 Days) as listed-below.

* Leeds Sleep Evaluation Questionnaire (LSEQ)
* Clinical examination - Scoring Based
* Sleep diary (sleeping time, the time interval in getting sleep, sleep interruptions, wake-up time, naps during the day, feeling, irritability, total duration of sleep, sleep quality.
* Product perception questionnaires (Product's effectiveness, likeliness and overall satisfaction- Hedonic scale (0-9-point scale)
* Blood parameter (CBC, ESR, RBS, SGOT, SGPT, S. Creatinine) - Safety Labs

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years (both inclusive) at the time of consent.
2. Sex: Healthy non-pregnant/non-lactating females and males.
3. Subject having difficulty in falling asleep due to shift work disturbance, jet lag, mental stress.
4. Female of childbearing potential must a reported negative pregnancy test, agree to follow an accepted method of birth control for the duration of the study such as condoms, foams, jellies, diaphragm, intrauterine device etc.
5. Subject is generally in good health.
6. Subjects who having > 30 minutes to fall asleep and subjective total sleep time of is 6.5 hours per night (for at least 3 nights per week); and daytime complaints associated with disturbed sleep.
7. Habitual bedtime between 8.30 pm to midnight.
8. Subject is willing to give written informed consent and are willing to follow the study procedure.
9. Agree to comply with all study procedures

Exclusion Criteria:

1. Subject has a history of allergy or sensitivity to the test treatment ingredients like melatonin, Tagar, minerals etc.
2. Subjects who suffer from sleep disorder other than primary insomnia including restless leg syndrome and sleep apnoea.
3. Subject who are substance dependence/ abuse in the past one year or with alcohol abuse.
4. Subject who are using tobacco products during night awakenings.
5. Subject with history of seizures or significant head trauma.
6. Subject worked on night or rotating shifts in previous 7 days before study initiation or who plan to do the same during the study period.
7. Subject Currently taking any medication on a regular basis (except for antihypertensives, antidiabetics, lipid lowering agents and drugs for primary cardiovascular prophylaxis).
8. Use of any:

   (i) Prescribed or over-the-counter (OTC) anti-inflammatory or medicine that leads to overweight like corticosteroids drugs within five (5) days prior to dosing.

   (ii) Antihistamine medication/immunosuppressive drugs within seven (7) days before first dosing.
9. Any other investigational drug was used within three months prior the entry in this study.
10. Subjects who cannot be relied upon to comply with the test procedures or are unwilling to give informed consent
11. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
12. Pregnant or breastfeeding or planning to become pregnant during the study period.
13. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials or skin care products within the last four weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of sleep | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms of change in quality of sleep by using Leed Sleep evaluation Questionnarie in which 0 indicate more difficult to 10 indicate Easier than usual
Change in duration sleep | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms of change in duration of sleep by using Leed Sleep evaluation Questionnarie in which 0 indicate more difficult to 10 indicate easier than usual

SECONDARY OUTCOMES:
Change in sleep quality by subjective self evaluated | From Day -7 (before usage) and Day 15 (post usage)
  To assess the effectiveness of test treatment in terms of change in sleep quality by using subjective Sleep diary
Improvement in overall health and wellbeing | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To assess the effectiveness of test treatment in terms Improvement in overall health and wellbeing by clinical examination
Subject product perception questionnaire | Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms of subject perception Questionnaire by using 9-point hedonic scale in which1 indicate extremely ineffective to 9 indicate extremely effective
Subject treatment perception | Day 30 (post usage)
  To evaluate the effectiveness of test treatment in terms dependence and withdrawal symptoms by telephonic follow up
Change in Complete Blood Count | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Complete Blood Count
Change in Erythrocyte Sedimentation Rate | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Erythrocyte Sedimentation Rate
Change in Random Blood Sugar | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Random Blood Sugar
Change in Serum Glutamate Pyruvate Transaminase | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Serum Glutamate Pyruvate Transaminase
Change in Serum Glutamate Oxaloacetic Transaminase | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Serum Glutamate Oxaloacetic Transaminase
Change in Serum Creatinine | From Baseline Day 01 (before usage) and Day 15 (post usage)
  To evaluate the effectiveness of test treatment in terms difference in Serum Creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No